CLINICAL TRIAL: NCT06124950
Title: A Couple-based Gender-transformative Intervention on Intimate Partner Violence Against Infertile Women
Brief Title: A Couple-based Gender-transformative Intervention on IPV Against Infertile Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Obstetrics and Gynecology Hospital (Other)
Responsible Party: Principal Investigator, Jie Qiao, Chief Physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: M2023460
Record Dates: First submitted 2023-10-20; First posted 2023-11-09 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Infertility, Female; Violence, Domestic
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GTI Intervention (Experimental): Participants in the intervention group will be provided with five GTI sessions (60-minutes/session) by trained nurses and social workers throughout participants' fertility treatment cycle throughout participants' fertility treatment cycle.
  Interventions: Behavioral: Gender-transformative intervention
- Standard Care (No Intervention): Participants in the intervention group will be provided with standard clinical procedures for assisted reproduction and health education.

INTERVENTIONS:
Behavioral: Gender-transformative intervention — A multidisciplinary team of experts, including 8-10 experts in reproductive medicine, nursing, social work, psychiatry, family law, and evidence-based medicine, will be established to support the development of the intervention.
  Five 60-minutes intervention sessions will be delivered by trained nurses and social workers throughout participants' fertility treatment cycle. Intervention will be carried out at the 5 critical windows of opportunity for infertility treatment: (1) before entering the cycle; (2) during follicular monitoring; (3) before oocyte retrieval; and (4) 2 weeks after the embryo transfer; and (5) 28-30 days after the embryo transfer.
  The intervention components will equip couples with educational information on health and relationship and skills obtained from interactive activities designed with an explicit focus on challenging gender stereotypes, all of which could incite reflection on sociocultural norms and gender-related power inequality.
  Arms: GTI Intervention

SUMMARY:
This is a multicenter, open-label, randomized controlled trial conducted at two reproductive medicine centers in Beijing, China. Couples undergoing their first or second in-vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) cycle, diagnosed with female-factor infertility, and who have signed informed consent will be enrolled. Exclusion criteria include couples receiving donated oocytes, sperm, or embryos; those diagnosed with severe male-factor infertility or unexplained infertility; those undergoing preimplantation genetic testing (PGT); those who have not undergone embryo transfer within six months after oocyte retrieval; those with severe mental disorders; and those who withdraw from the study.

Participants are will randomly allocated 1:1 by center to either the intervention or control group. Couples in the intervention group will receive five 60-minutes GTI sessions focusing on gender norms, gender equality, and healthy relationship skills, conducted by trained healthcare providers and social workers. The control group will receive standard reproductive care. A total of 376 infertile couples will be enrolled (188 couples per group).

The primary outcome is the IPV rate against infertile women over the past 12 months.

DETAILED DESCRIPTION:
Infertility and intimate partner violence (IPV) are significant challenges in sexual and reproductive health, with a notable intersection as infertile women face higher IPV risks. However, the needs of infertile couples have been largely overlooked, and the effectiveness of gender-transformative interventions (GTIs) designed to challenge gender inequality and question gender norms in reducing IPV against infertile women has not been evaluated.

This is a multicenter, open-label, randomized controlled trial conducted at two reproductive medicine centers in Beijing, China (the Centers for Reproductive Medicine of Peking University Third Hospital and Beijing Obstetrics and Gynecology Hospital).

A multidisciplinary team of experts, including 8-10 experts in reproductive medicine, nursing, social work, psychiatry, family law, and evidence-based medicine, will be established to support the development of the intervention. Five 60-minutes GTI sessions will be delivered by trained nurses and social workers throughout participants' fertility treatment cycle. Intervention will be carried out at the 4 critical windows of opportunity for infertility treatment: (1) before entering the cycle; (2) during follicular monitoring; (3) the oocyte retrieval-embryo transfer phase; (4) 2 weeks after the embryo transfer (hCG pregnancy test), and (5) 28-30 days after the embryo transfer. The intervention components will equip couples with educational information on health and relationship and skills obtained from interactive activities designed with an explicit focus on challenging gender stereotypes, all of which could incite reflection on sociocultural norms and gender-related power inequality.

Participants are will randomly allocated 1:1 by center to either the intervention or control group. Couples in the intervention group will receive GTI sessions. The control group will receive standard reproductive care. A total of 376 infertile couples will be enrolled (188 couples per group).

ELIGIBILITY:
Inclusion Criteria:

* Couples who are undergoing their first or second IVF/ICSI cycle;
* Couples diagnosed with female-factor infertility;
* Couples who have signed consent.

Exclusion Criteria:

* Couples who receive donated oocytes, sperm, or embryos;
* Couples diagnosed with severe male-factor infertility or unexplained infertility.
* Couples who are undergoing Preimplantation Genetic Testing (PGT);
* Couples who have not undergone embryo transfer within six months after oocyte retrieval;
* Couples who have severe mental disorders;
* Couples who withdrew from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Past-12-months Intimate Partner Violence against infertile women | T0 (Baseline) and T0 + ~14 months (4 weeks after delivery)
  Past-12-months prevalence of IPV against infertile women measured using an instrument that combined the Revised Conflict Tactics Scale (CTS-2) and the Scale of Economic Abuse-12 (SEA-12).
  Respondents will be asked if they had experienced any specific acts of physical (6 items from CTS-2 injury subscale, 12 from CTS-2 physical assault subscale), psychological (8 items from CTS-2 psychological aggression subscale), sexual (7 items from CTS-2 sexual coercion subscale), or economic violence (12 items from SEA-12) in the past 12 months.
  The past-12-months prevalence of IPV is calculated as the proportion of participants reporting at least one act of violence in the past 12 months.

SECONDARY OUTCOMES:
Past-12-months Intimate Partner Violence against male partners | T0 (Baseline) and T0 + ~14 months (4 weeks after delivery)
  Past-12-months prevalence of IPV against male partners measured using an instrument that combined the Revised Conflict Tactics Scale (CTS-2) and the Scale of Economic Abuse-12 (SEA-12).
  Respondents will be asked if they had experienced any specific acts of physical (6 items from CTS-2 injury subscale, 12 from CTS-2 physical assault subscale), psychological (8 items from CTS-2 psychological aggression subscale), sexual (7 items from CTS-2 sexual coercion subscale), or economic violence (12 items from SEA-12) in the past 12 months.
  The past-12-months prevalence of IPV is calculated as the proportion of participants reporting at least one act of violence in the past 12 months.
Past-3-months Intimate Partner Violence against infertile women | T0 (Baseline); T0 + ~2months (28-30 days after embryo transfer); T0 + ~4 months (12-13 weeks of gestation); T0 + ~12-14 months (4 weeks after delivery)
  Past-3-months prevalence of IPV against infertile women measured using the World Health Organization Violence Against Women (WHO-VAW) Instrument.
  The WHO-VAW has 6 items asking if participants had experienced any specific acts of physical (1 item), sexual (1 item), and psychological (4 items) violence in the past 3 months.
  The past-3-months prevalence of IPV is calculated as the proportion of participants reporting at least one act of violence in the past 3 months.
Past-3-months Intimate Partner Violence against male partners | T0 (Baseline); T0 + ~2months (28-30 days after embryo transfer); T0 + ~4 months (12-13 weeks of gestation); T0 + ~12-14 months (4 weeks after delivery)
  Past-3-months prevalence of IPV against male partners measured using the World Health Organization Violence Against Women (WHO-VAW) Instrument.
  The WHO-VAW has 6 items asking if participants had experienced any specific acts of physical (1 item), sexual (1 item), and psychological (4 items) violence in the past 3 months.
  The past-3-months prevalence of IPV is calculated as the proportion of participants reporting at least one act of violence in the past 3 months.
Past-12-months Severe Intimate Partner Violence against infertile women | T0 (Baseline) and T0 + ~14 months (4 weeks after delivery)
  Past-12-months prevalence of severe IPV against infertile women measured using an instrument that combined the Revised Conflict Tactics Scale (CTS-2) and the Scale of Economic Abuse-12 (SEA-12).
  Respondents will be asked if they had experienced any specific acts of physical (6 items from CTS-2 injury subscale, 12 from CTS-2 physical assault subscale), psychological (8 items from CTS-2 psychological aggression subscale), sexual (7 items from CTS-2 sexual coercion subscale), or economic violence (12 items from SEA-12) in the past 12 months.
  Severe IPV is defined as any reported instance of physical or sexual violence (regardless of frequency) and/or any psychological or economic violence ≥ 3 times in the past year.
  The past-12-months prevalence of severe IPV is calculated as the proportion of participants reporting at least one severe IPV in the past 12 months.
Past-12-months severe Intimate Partner Violence against male partners | T0 (Baseline) and T0 + ~14 months (4 weeks after delivery)
  Past-12-months prevalence of severe IPV against male partners measured using an instrument that combined the Revised Conflict Tactics Scale (CTS-2) and the Scale of Economic Abuse-12 (SEA-12).
  Respondents will be asked if they had experienced any specific acts of physical (6 items from CTS-2 injury subscale, 12 from CTS-2 physical assault subscale), psychological (8 items from CTS-2 psychological aggression subscale), sexual (7 items from CTS-2 sexual coercion subscale), or economic violence (12 items from SEA-12) in the past 12 months.
  Severe IPV is defined as any reported instance of physical or sexual violence (regardless of frequency) and/or any psychological or economic violence ≥ 3 times in the past year.
  The past-12-months prevalence of severe IPV is calculated as the proportion of participants reporting at least one severe IPV in the past 12 months.
Attitudes toward male gender roles | T0 (Baseline); T0 + ~2months (28-30 days after embryo transfer); T0 + ~4 months (12-13 weeks of gestation); T0 + ~12-14 months (4 weeks after delivery)
  Attitudes toward male gender roles measured by the Male Role Attitudes Scale (MRAS) to assess infertile couples' attitudes towards traditional male role stereotypes.
  The MRAS has 8 items. Responses to the MRAS were based on a four-point Likert scale from 'strongly disagree=1' to 'strongly agree=4'. A total score was derived by totalling responses to each item, giving a possible score of 8-32, where higher scores indicate greater endorsement of traditional male role stereotypes.
Martial quality and satisfaction | T0 (Baseline); T0 + ~2months (28-30 days after embryo transfer); T0 + ~4 months (12-13 weeks of gestation); T0 + ~12-14 months (4 weeks after delivery)
  Martial quality and satisfaction measured by the Relationship Assessment Scale (RAS).
  The RAS has 7 items. Responses to the RAS were based on a five-point Likert scale from 'low=1' to 'high=5'. Items 4 and 7 are reverse-scored. A total score was derived by totalling responses to each item, giving a possible score of 7-35. The higher the score, the more satisfied the respondent is with his/her relationship.
Couples' coping with stress | T0 (Baseline); T0 + ~2months (28-30 days after embryo transfer); T0 + ~4 months (12-13 weeks of gestation); T0 + ~12-14 months (4 weeks after delivery)
  Couples' coping with stress was measured by two items from the Dyadic Coping Inventory (DCI).
  Responses to the DCI were based on a five-point Likert scale ranging from 'strongly disagree = 1' to 'strongly agree = 5'.A total score was derived by totalling responses to each item, giving a possible score of 2-10. A higher score indicates couple's better dyadic coping with stress.
Patient satisfaction with infertility treatment | T0 (Baseline); T0 + ~2months (28-30 days after embryo transfer); T0 + ~4 months (12-13 weeks of gestation); T0 + ~12-14 months (4 weeks after delivery)
  Patient satisfaction was measured by one item from the patient satisfaction survey.
  Responses to this question were based on a five-point Likert scale ranging from 'strongly disagree = 1' to 'strongly agree = 5'. The score ranged from 1 to 5, with a higher score indicating greater satisfaction with the infertility treatment.
Human chorionic gonadotropin (hCG) Positive | T0 + ~1.5 months
  Positive for Beta-human chorionic gonadotropin (βhCG) in blood or urine after embryo transfer.
Clinical pregnancy | T0 + ~2 months (28-30 days after embryo transfer)
  One or more observed gestational sac or definitive clinical signs of pregnancy under ultrasonography at 28-30 days after embryo transfer (including clinically documented ectopic pregnancy).
Ongoing pregnancy | T0 + ~4 months (12 weeks after embryo transfer)
  Presence of a gestational sac and fetal heartbeat after 12 weeks of gestation.
Miscarriage | 22 weeks of gestation
  Spontaneous loss of an intra-uterine pregnancy prior to 22 completed weeks of gestational age.
Biochemical Pregnancy Loss | T0 + 1.5-2 months
  Positive for hCG after embryo transfer, but no clinical pregnancy observed.
Stillbirth | After 22 weeks of gestation
  Fetal death after 22 weeks of gestation, with no signs of life such as heartbeat, breathing, umbilical cord pulse, or voluntary muscle contraction.
Live birth | After 22 weeks of gestation
  A delivery of one or more living infants (≥22 weeks gestation or birth weight more than 1,000g).
Ectopic pregnancy | 7 weeks of gestation
  Implantation takes place outside the uterine cavity, confirmed by sonography or laparoscopy.
Cycle cancellation | T0 + ~2 months
  The cycle is considered canceled if any of the following situations occur from the ovarian stimulation to the embryo transfer:
  1. The researcher determines that by the 20th day of ovarian stimulation, there are not ≥2 follicles with a diameter of ≥18mm.
  2. Ultrasound reveals more than 25 follicles with a diameter of ≥12mm.
  3. No oocytes are retrieved on the egg retrieval day.
  4. No transferable embryos are available on the transfer day.
  5. Ovarian Hyperstimulation Syndrome (OHSS) occurs during the ovarian stimulation process.
  6. The participant requests to cancel the cycle or the researcher cancels the cycle for other valid reasons.
Preterm birth | 28-37 weeks of pregnancy
  Birth of a fetus delivered after 28 and before 37 completed weeks of gestational age in participants confirmed ongoing pregnancy.
Birth weight | Within the first hour after live birth
  The weight measured for the first time within the first hour after birth. High birth weight: ≥4kg; Low birth weight: < 2.5kg.
Congenital anomaly | Within 2 weeks after live birth
  Any congenital anomaly will be included, including structural or chromosomal abnormalities of the fetus in utero, Trisomy 21 (Down syndrome), congenital heart disease, neural tube defects, cleft lip and palate, polydactyly, hydrocephalus, etc.
Neonatal mortality | Within 28 days of birth
  Death of a live born baby within 28 days of birth

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, Dr, Principal Investigator — Peking University Third Hospital
Locations (2):
- China (2):
  - Beijing Obstetrics and Gynecology Hospital, Beijing
  - Peking University Third Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No
Given the nature of the study, individual participant data (IPD) will not be available to other researchers.